CLINICAL TRIAL: NCT02105038
Title: Effects of Upper Extremity Immobilization and Use of a Steering Wheel Spinner Knob Following Distal Radius Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: Pro00026777
Record Dates: First submitted 2014-03-24; First posted 2014-04-07 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Distal Radius Fracture
Keywords: distal radius fracture; steering; steering wheel spinner knob
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Knob (Experimental): Steering in a driving simulator using a steering wheel spinner knob.
  Interventions: Other: Spinner knob
- No Knob (Active Comparator): Steering in a driving simulator immediately following surgical treatment of hip fractures.
  Interventions: Other: No Knob

INTERVENTIONS:
Other: Spinner knob
  Arms: Knob
Other: No Knob
  Arms: No Knob

SUMMARY:
The aims of the study are to better understand how upper extremity injury and immobilization influences a patient's steering ability. Patients with acute distal radius fractures treated with surgery will be recruited for study in a driving simulator. The results will hopefully assist physicians to better counsel patients with upper extremity injuries on when it is safe to return to driving.

DETAILED DESCRIPTION:
The ability of an injured person to safely drive an automobile while immobilized in an upper extremity cast or splint is not well defined.

The aims of the study are to better understand how upper extremity injury and immobilization influences a patient's steering ability. The secondary aim is to further evaluate the effectiveness of a steering wheel spinner-knob to assist with one-handed driving. A steering wheel spinner knob may be a surrogate to assist with one handed driving while immobilized.

ELIGIBILITY:
Inclusion Criteria:

* • Acute distal radius fracture treated with surgery and initially immobilized in a cast or splint

  * Valid driver's license with 1 years of driving experience and actively driving during the last three months
  * English speaking
  * Ability to start testing within 10 days of surgery

Exclusion Criteria:

* • <18 years of age

  * Current use of steering wheel spinner knob or hand controls while driving
  * Non-drivers
  * Multi-trauma
  * Open fractures
  * Surgical repair with external fixation
  * Concurrent distal radius/ulnar joint injury and repair
  * Any other joint besides the wrist immobilized following surgery
  * Contralateral upper extremity disability
  * Previous ipsilateral upper extremity functional deficit
  * Inability to participate for the full length of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Steering reaction time | 6 months
  Steering reaction time measured using a driving simulator will be compared across three time points (acutely, sub-acutely, and return to function) following surgical treatment of a distal radius fractures. This will be evaluated with and without the use of a steering wheel spinner knob.

SECONDARY OUTCOMES:
Steering accuracy | 6 months
  Steering accuracy measured using a driving simulator will be compared across three time points (acutely, sub-acutely, and return to function) following surgical treatment of a distal radius fractures. This will be evaluated with and without the use of a steering wheel spinner knob.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle J Jeray, MD, Principal Investigator — Prisma Health-Upstate
Locations (1):
- Greenville Health System, Greenville, South Carolina, United States